CLINICAL TRIAL: NCT05962918
Title: The Effects of Perineal Massage Performed During Labor on Childbirth Comfort, Perineal Pain and Trauma in Nulliparous Women: A Quasi Experimental Study
Brief Title: Perineal Massage Performed During the Labour
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Munzur University (Other)
Responsible Party: Principal Investigator, Habibe YAŞAR YETİŞMİŞ, Research assistant, Phd Student, Munzur University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: habibe4721
Record Dates: First submitted 2023-05-31; First posted 2023-07-27 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Delivery Problem; Childrearing; Satisfaction, Patient; Perineum; Injury; Perineal Tear; Pain, Labor
Keywords: Childbirth comfort; Perineal massage; Perineal tear; Perineal pain; midwifery
MeSH Terms: conditions — Dystocia; Patient Satisfaction; Wounds and Injuries; Labor Pain

STUDY DESIGN:
Intervention Model Description: Paralel designed non randomized two armed study
Who Masked: Participant
Masking Description: Since the researcher did the intervention and analysis, only the participants did not know which group they were in, so single blinding was done.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- perineal massage (Experimental): intervention group with perineal massage
  Interventions: Other: Perinal massage
- control group (No Intervention): The group that received routine hospital protocol and was not massaged.

INTERVENTIONS:
Other: Perinal massage — Perineal massage was administered to all pregnant women in the experimental group during both the labor and resting phases between contractions. The participants received an average of 5-10 minutes of perineal massage two, four and four to six times at the latent (0-3-cm cervical dilation), active (4-7-cm cervical dilation) and transition (8-10-cm cervical dilation) phases of labor, respectively. These women continued to receive perineal massage at every push throughout the second stage of labor. The researcher midwife gently widened the perineal muscles by making stretching movements with her fingers. Perineal massage was applied using all three of the "from one edge to the other", "U shape" and "pressure" massage techniques. The researcher gently applied a rhythmic "U" pressure with both fingers, moving them on the vagina downwards about 3 to 9 o'clock. Each pressure movement was maintained laterally for 1-2 minutes towards the rectum.
  Arms: perineal massage

SUMMARY:
In this study, perineal massage was applied to primiparous women who did not give birth before, as a quasi-experimental control group to determine the effects of massage on birth comfort, perineal trauma and perineal pain.

DETAILED DESCRIPTION:
In this study, perineal massage was applied to primiparous women who did not give birth before, as a quasi-experimental control group to determine the effects of massage on birth comfort, perineal trauma and perineal pain. Perineal massage was administered to all pregnant women in the experimental group during both the labor and resting phases between contractions. The participants received an average of 5-10 minutes of perineal massage two, four and four to six times at the latent (0-3-cm cervical dilation), active (4-7-cm cervical dilation) and transition (8-10-cm cervical dilation) phases of labor, respectively. These women continued to receive perineal massage at every push throughout the second stage of labor. Before perineal massage, the researcher wore sterile gloves, placed two fingers into the 3-4-cm wide-open vagina and applied Vaseline routinely to lubricate the vagina in the delivery room. . Perineal massage was applied using all three of the "from one edge to the other", "U shape" and "pressure" massage techniques. The researcher gently applied a rhythmic "U" pressure with both fingers, moving them on the vagina downwards about 3 to 9 o'clock. Each pressure movement was maintained laterally for 1-2 minutes towards the rectum.

ELIGIBILITY:
Inclusion Criteria:

* Having no complications for vaginal delivery
* Having no dystocia affecting the birth process (e.g., prolonged labor, precipitate labor, shoulder dystocia)
* Having a singleton pregnancy,
* Having a fetal head with an anterior cephalic position,
* Being at the latent phase of labor,
* Having no perineal scar tissue,
* Having no diagnosis of vaginal fungus or infection,
* Having a fetus with a birth weight between 2500 and 4000 g,
* Having no communication problems.

Exclusion Criteria:

-All pregnant women who developed fetal distress during labor or had to undergo cesarean delivery were excluded from the study.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 182 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
Change in perineal pain scores | 4-6 hours after the childbirth
  The mean visual analog scale (VAS) scores of the pregnant women in the experimental and control groups were compared to determine the level of perineal pain. Women were asked to rate pain from zero to 10. A score of zero means no pain, while 10 = indicates the most severe pain experienced.
Change in childbirth comfort scores | 4-6 hours after coming to labor
  The "Childbirth Comfort Questionnaire (CCQ)" score averages were compared to determine the birth comfort levels of the pregnant women in the experimental and control groups. As the score increases, high-level comfort is mentioned, as the score decreases, low-level comfort is mentioned. The lowest and highest possible total scale scores are 9 and 45.
Change in perineal trauma scores | 4-6 hours after the childbirth.
  The REEDA scale mean scores were compared to determine the perineal trauma levels of the women in the experimental and control groups. The REEDA scale, consists of five variables of wound healing. These variables are redness, edema, ecchymosis, discharge and approximation of the wound edges. The scale items are scored between 0 and 3 points. The lowest and highest possible total scale scores are 0 and 15. A higher score indicates a greater level of perineal trauma.

CONTACTS AND LOCATIONS:
Locations (1):
- Munzur University, Tunceli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Labrecque M, Eason E, Marcoux S, Lemieux F, Pinault JJ, Feldman P, Laperriere L. Randomized controlled trial of prevention of perineal trauma by perineal massage during pregnancy. Am J Obstet Gynecol. 1999 Mar;180(3 Pt 1):593-600. doi: 10.1016/s0002-9378(99)70260-7. PMID 10076134
- [Background] Aquino CI, Guida M, Saccone G, Cruz Y, Vitagliano A, Zullo F, Berghella V. Perineal massage during labor: a systematic review and meta-analysis of randomized controlled trials. J Matern Fetal Neonatal Med. 2020 Mar;33(6):1051-1063. doi: 10.1080/14767058.2018.1512574. Epub 2018 Sep 19. PMID 30107756
- [Background] Karacam Z, Ekmen H, Calisir H. The use of perineal massage in the second stage of labor and follow-up of postpartum perineal outcomes. Health Care Women Int. 2012;33(8):697-718. doi: 10.1080/07399332.2012.655385. PMID 22827728
- [Background] Williams A, Herron-Marx S, Knibb R. The prevalence of enduring postnatal perineal morbidity and its relationship to type of birth and birth risk factors. J Clin Nurs. 2007 Mar;16(3):549-61. doi: 10.1111/j.1365-2702.2006.01593.x. PMID 17335531
- [Background] Kalichman L. Perineal massage to prevent perineal trauma in childbirth. Isr Med Assoc J. 2008 Jul;10(7):531-3. No abstract available. PMID 18751635
- [Background] Geranmayeh M, Rezaei Habibabadi Z, Fallahkish B, Farahani MA, Khakbazan Z, Mehran A. Reducing perineal trauma through perineal massage with vaseline in second stage of labor. Arch Gynecol Obstet. 2012 Jan;285(1):77-81. doi: 10.1007/s00404-011-1919-5. Epub 2011 May 26. PMID 21614497
- [Result] Akhlaghi F, Sabeti Baygi Z, Miri M, Najaf Najafi M. Effect of Perineal Massage on the Rate of Episiotomy. J Family Reprod Health. 2019 Sep;13(3):160-166. PMID 32201491
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/29238501/